CLINICAL TRIAL: NCT00991757
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of RWJ 333369 as Adjunctive Therapy in Subjects With Partial Onset Seizures Followed by an Open-Label Extension Study: Open-Label Extension Period
Brief Title: An Open-Label Extension Study to Evaluate the Safety and Tolerability of RWJ 333369 as Adjunctive Therapy in Patients 16 Years and Older With Partial Onset Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 333369EPY3004
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Epilepsy; Complex Partial Seizures; Epilepsy, Complex Partial; Epilepsies, Partial
Keywords: RWJ-333369; Anticonvulsants; Antiepileptic drugs; Epilepsy, Focal; Seizure Disorder
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsy, Complex Partial; Epilepsies, Partial | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

ARMS (1):
- 001 (Experimental): carisbamate Open-Label Extension: 400 mg/day (up to a maximum of 1200mg/day) given in 2 equally divided doses for up to 1 year (or until carisbamate is available by prescription or the sponsor terminates the study).
  Interventions: Drug: carisbamate

INTERVENTIONS:
Drug: carisbamate — Open-Label Extension: 400 mg/day (up to a maximum of 1200mg/day) given in 2 equally divided doses for up to 1 year (or until carisbamate is available by prescription or the sponsor terminates the study).

SUMMARY:
The purpose of this open-label extension study is to demonstrate that RWJ-333369 is safe as long-term add-on treatment of partial onset seizures.

DETAILED DESCRIPTION:
333369EPY3004 is the open-label extension study that follows the double-blind studies 333369EPY3001 and 333369EPY3002 (NCT00425282 and NCT00433667, respectively). In an open label study such as 333369EPY3004, both the physician and the patient know the name of the assigned study medication. In a double blind study such as 333369EPY3001 and 333369EPY3002, neither the physician nor the patient knows the name of the assigned study medication. Patients who complete the double-blind treatment phase of studies 333369EPY3001 and 333369EPY3002 will be eligible to enter the open-label extension study 333369EPY3004 during which patients will transition through a blinded period to an open-label period with carisbamate (also referred to as RWJ-333369). There will be a blinded transition during which patients will take blinded study medication; after this, patients will then take unblinded, open-label study medication. No patients will receive placebo during the open-label extension. Safety assessments include the monitoring of the frequency, severity, and timing of adverse events, clinical laboratory test results, 12-lead electrocardiogram (ECG) recordings, vital signs measurements, physical and neurologic examinations, the Physician Withdrawal Checklist for symptoms of withdrawal for those patients who taper and/or discontinue study drug, and pregnancy tests for females of childbearing potential. Seizure counts will be obtained at every visit. A Quality of Life in Epilepsy questionnaire will be administered during the study. There is no statistical testing hypothesis for this study. Detailed Description update,5 Oct 2009. The Sponsor in conjunction with the DSMB agreed to amend the protocol to withdraw patients who develop signs of a drug hypersensitivity reaction. Open-label treatment with carisbamate 400 mg/day (up to a maximum of 1200mg/day) given in 2 equally divided doses BID for up to 1 year; study drug should be swallowed whole and not be chewed, divided, crushed, or dissolved.

ELIGIBILITY:
Inclusion Criteria:

* In order to enter the open label extension, the patient must have completed either Study 333369EPY3001 or Study 333369EPY3002.

Exclusion Criteria:

* Generalized epilepsy
* Currently experiencing seizures that cannot be counted accurately
* Unstable medical disease, such as a recent heart attack or uncontrolled diabetes
* Major psychiatric illness
* Recent drug or alcohol abuse
* Unable to swallow pills

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 991 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Worsening of seizures, including rates of status epilepticus. | Up to approximately 48 months

SECONDARY OUTCOMES:
Quality of Life in Epilepsy-31-Problems (QOLIE-31-P) | month 6

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.